CLINICAL TRIAL: NCT03977194
Title: Phase III Randomized Trial of Atezolizumab in Elderly Patients With Advanced Non-Small-Cell Lung Cancer and Receiving Monthly Carboplatin With Weekly Paclitaxel Chemotherapy
Brief Title: Atezolizumab in Elderly Patients With Advanced Non-Small-Cell Lung Cancer and Receiving Carboplatin Paclitaxel Chemotherapy
Acronym: ELDERLY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1805
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: IFCT; ELDERLY; NSCLC; immunotherapy; chemotherapy
MeSH Terms: interventions — Carboplatin; Paclitaxel; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : standard treatment (Active Comparator): Carboplatine + paclitaxel (4 cycles of 28 days)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Arm B : standard treatment + immunotherapy (Experimental): Carboplatine + paclitaxel (4 cycles of 28 days) + atezolizumab (every 21 days) until progression or toxicity
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Atezolizumab

INTERVENTIONS:
Drug: Carboplatin — AUC 6 every 4 weeks
Drug: Paclitaxel — 90 mg/m² D1, 8, 15, every 4 weeks
Drug: Atezolizumab — 1200 mg every 3 weeks
  Arms: Arm B : standard treatment + immunotherapy

SUMMARY:
Non Small Cell Lung Cancer (NSCLC) remains the leading cause of death by cancer in the world. Because of the increase in lung cancer incidence with age and the increase of life expectancy, about half of the patients are patients aged 70 or older. Several clinical trials have shown the interest of adding immunotherapy to standard 1st line chemotherapy in NSCLC. Although in these studies there was not necessarily a higher age limit, in fact the proportion of included patients aged 75 or older remains low (between 7 and 10%). It is therefore necessary to conduct a trial dedicated to these patients in order to determine whether immunotherapy is as effective and tolerated as in the general population.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent:

   * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing
2. Histologically confirmed NSCLC. A cytologically-proven NSCLC is allowed if a cytoblock has been prepared.
3. Age: 70 to 89 years
4. Performance status ≤1.
5. Stage IIIB or IIIC non irradiable or IV (8th classification TNM, UICC 2015)
6. Measurable disease as defined by RECIST 1.1. The radiological assessment has to be done within the timelines indicated.
7. No prior systemic anticancer therapy (including EGFR or ALK inhibitors) given as primary therapy for advanced or metastatic disease. Previously irradiated lesion must not be the only measurable site of disease.
8. At least 3 weeks must have elapsed after major surgery or radiation therapy
9. Adequate biological functions:

   Creatinine Clearance ≥ 45 mL/min (Cockcroft or MDRD or CKD-epi); neutrophiles ≥ 1500/mm3 ; platelets ≥100 000/mm3 ; Hemoglobin ≥ 9g/dL ; hepatic enzymes < 3x ULN except for patients with hepatic metastases (< 5 x ULN), total bilirubin ≤ 1,5 x ULN except for patients with proved, Gilbert syndrome (≤ 5 x ULN) or patients with hepatic metastases (≤ 3,0 mg/dL).
10. Life expectancy of at least 12 weeks
11. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 6 months after the last dose of treatment. Male patients should not donate sperm during this study and for at least 6 months after the last dose of treatment.

    Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the treatment. Male patients must always use a condom.
12. Patient covered by a national health insurance
13. Protected adults can participate if they are able to make decision about their medical treatment according to guardianship judgment.

Exclusion Criteria:

1. Small cell lung cancer or tumors with mixt histology including a SCLC component
2. Known EGFR activating tumor mutation.
3. Known ALK or ROS1 gene rearrangement as assessed by IH, FISH or NGS sequencing
4. Previous or active cancer within the previous 3 years with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal cell skin cancer or ductal carcinoma in situ treated surgically with curative intent. For other type of cancer, please contact IFCT). Patients with a prostate adenocarcinoma history within the previous 3 years could be included in case of localized prostate cancer, with good prognostic factors according to d'Amico classification (≤ T2a and Score de Gleason ≤ 6 and PSA (ng/ml) ≤ 10), provided they were treated in a curative way (surgery or radiotherapy ± hormonotherapy, without any chemotherapy)
5. Mini Mental Score < 24
6. Previous systemic treatment (including but not limited to chemotherapy, targeted treatment or immunotherapy) except for adjuvant therapy given more than 5 years ago.
7. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
8. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
9. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.

   Patients with rheumatoid arthritis without exacerbation during one year and with no more than 10 mg oral prednisone /day or equivalent may be included after rheumatologist advice.

   Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin regimen are eligible for this study

   Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
   * Rash must cover less than 10% of body surface area (BSA).
   * Disease is well controlled at baseline and only requiring low potency topical steroids.
   * No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
10. Symptomatic brain metastases requiring corticosteroids.
11. Spinal cord compression not definitely treated by surgery and/or radiation therapy or with neurological sequelae.
12. Leptomeningeal disease
13. Uncontrolled tumor-related pain.
14. Uncontrolled or symptomatic or requiring Denosumab hypercalcemia .
15. Corticosteroids > 10mg oral prednisone/day or equivalent.
16. Immunosuppressive medications within 2 weeks before randomization
17. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
18. HIV positive serology (test at screening),
19. Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen HBsAg test at screening) or hepatitis C Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible only if they are negative for HBV DNA.

    Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
20. Active tuberculosis
21. Severe infection within 4 weeks before randomization
22. Received therapeutic oral or iv antibiotics within 2 weeks before randomization.
23. Administration of live attenuated vaccine within four weeks before randomization or anticipation that such a live attenuated vaccine will be required during the study.
24. Serious undergoing diseases or comorbidities precluding the possibility for the patient to receive the treatments, including but not limited to unstable angina or uncontrolled cardiac disease.
25. Polyneuropathy ≥ grade 2 CTC
26. Treatment with an investigational drug during the 4 weeks preceding inclusion in the trial.
27. Known allergy to Cremophor EL

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 510 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 11 months after randomization of the last subject
  Time from randomization until death due to any cause

SECONDARY OUTCOMES:
Progression-free survival | 11 months after randomization of the last subject
  Time from randomization to first observation of progression (according to RECIST v1.1) or date of death (from any cause).
Best overall response rate | 11 months after randomization of the last subject
  Best response according to RECIST v1.1 from start to end of study treatment
Duration of response | 11 months after randomization of the last subject
  Time from documentation of tumor response to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth QUOIX, Study Chair — Strasbourg - NHC; Céline MASCAUX, Study Chair — Strasbourg - NHC
Locations (68):
- France (68):
  - Abbeville - CH, Abbeville
  - Aix-en-Provence - CH, Aix-en-Provence
  - Annemasse - CH, Ambilly
  - Metz - Thionville CHR, Ars-Laquenexy
  - Auxerre - CH, Auxerre
  - Avignon - Institut Sainte-Catherine, Avignon
  - Avignon - CH, Avignon
  - Bayonne - CH, Bayonne
  - Besançon - CHU, Besançon
  - Bobigny - APHP - Hôpital Avicenne, Bobigny
  - Bordeaux - CHU Hôpital Haut-Lévèque, Bordeaux
  - Bordeaux - Polyclinique Nord, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne-Billancourt
  - Caen - CHU Côte de Nacre, Caen
  - Cannes - CH, Cannes
  - Carcassone - CH, Carcassonne
  - Centre Hospitalier de Chambéry, Chambéry
  - Chauny - Centre Hospitalier, Chauny
  - Cholet - CH, Cholet
  - Clamart - Hôpital Percy, Clamart
  - Clermont Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Cornebarrieu - Clinique des Cèdres, Cornebarrieu
  - Dijon - Centre Georges-François Leclerc, Dijon
  - Grenoble - CHU, Grenoble
  - Le Mans - CHG, Le Mans
  - Lille - GHICL, Lille
  - Lille - Polyclinique de la Louvière, Lille
  - Limoges - CHU, Limoges
  - Lorient - CHBS, Lorient
  - Lyon - Hôpital Jean Mermoz, Lyon
  - Marseille - AP-HM Hôpital Nord, Marseille
  - Marseille - Hôpital Européen, Marseille
  - Marseille - Institut Paoli Calmette, Marseille
  - Meaux - CH, Meaux
  - Montauban - CH, Montauban
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - Mulhouse - GHRMSA, Mulhouse
  - Nancy - Institut de Cancérologie de Lorraine, Nancy
  - Nantes - CHU Hôpital Laënnec, Nantes
  - Nice - CRLCC, Nice
  - Orléans - CH, Orléans
  - Paris - Hôpital Saint Joseph, Paris
  - Paris - APHP - Hopital Tenon, Paris
  - Paris - APHP Bichat, Paris
  - Paris - Curie, Paris
  - Paris - Hôpital Cochin, Paris
  - Pau - CHG, Pau
  - Lyon - URCOT, Pierre-Bénite
  - Quint-Fonsegrives - Clinique de la Croix du Sud, Quint-Fonsegrives
  - Rodez - CH, Rodez
  - Saint-Cloud - Centre René Huguenin, Saint-Cloud
  - La Réunion - CHU (site Félix GUYON), Saint-Denis
  - Saint-Etienne - CHU, Saint-Etienne
  - Centre Hospitalier Mémorial de Saint-Lô, Saint-Lô
  - Saint- Mandé - HIA Begin, Saint-Mandé
  - La Réunion - CHU (Site Sud), Saint-Pierre
  - Saint-Priest - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Sens - CH, Sens
  - Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Toulon - CHI, Toulon
  - Toulon - HIA, Toulon
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
  - Valence - CH, Valence
  - Valenciennes - Clinique, Valenciennes
  - Villefranche-Sur-Saône - Hôpital Nord-Ouest, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data underlying the results reported in this article, as well as the study protocol and statistical analysis plan, will be made available after deidentification immediately following publication and for three years. Researchers who provide a methodologically sound proposal for any purpose may direct proposals to contact@ifct.fr. To gain access, data requestors will need to sign a data access agreement that requires approval by the French Cooperative Thoracic Intergroup.

REFERENCES:
- [Background] Quoix E, Zalcman G, Oster JP, Westeel V, Pichon E, Lavole A, Dauba J, Debieuvre D, Souquet PJ, Bigay-Game L, Dansin E, Poudenx M, Molinier O, Vaylet F, Moro-Sibilot D, Herman D, Bennouna J, Tredaniel J, Ducolone A, Lebitasy MP, Baudrin L, Laporte S, Milleron B; Intergroupe Francophone de Cancerologie Thoracique. Carboplatin and weekly paclitaxel doublet chemotherapy compared with monotherapy in elderly patients with advanced non-small-cell lung cancer: IFCT-0501 randomised, phase 3 trial. Lancet. 2011 Sep 17;378(9796):1079-88. doi: 10.1016/S0140-6736(11)60780-0. Epub 2011 Aug 8. PMID 21831418
- See also: IFCT website — https://www.ifct.fr/index.php/fr/la-recherche/item/2149-ifct-1805-elderly